CLINICAL TRIAL: NCT02635932
Title: Effectiveness of Trapeziometacarpal Splint
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Fabiana de Carvalho Silva, Physiotherapist, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEP_UNIFESP_269.012
Record Dates: First submitted 2015-12-13; First posted 2015-12-21 (Estimated); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Osteoarthritis of Trapeziometacarpal Joint

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Functional Splint group (Experimental): Patient will be using the functional splint during their activity daily life
  Interventions: Device: Day Splint
- Night Splint group (Active Comparator): Patients will use the night splint during the sleep time
  Interventions: Device: Night Splint

INTERVENTIONS:
Device: Day Splint — A thermoplastic splint was confected for each participant to stabilize the trapeziometacarpal joint, maintaining the pulp of the distal phalange of the index finger free for gripping with the other fingers and leaving the thumb in a functional position. In this group the slint was used during the daily life activities.
  Arms: Functional Splint group
Device: Night Splint — A thermoplastic splint was confected for each participant to stabilize the trapeziometacarpal joint, maintaining the pulp of the distal phalange of the index finger free for gripping with the other fingers and leaving the thumb in a functional position. In this group the slint was used during the night.
  Arms: Night Splint group

SUMMARY:
The trapeziometacarpal osteoarthritis is a degenerative or inflammatory joint that affects the trapeziometacarpal joint (TMC) of the thumb. Its main symptom is pain that leads to difficulty in manual function and decrease the patient's quality of life. Immobilization of TMC thumb joint by bracing has been effective in reducing pain and improving function. Objective: To compare the effectiveness between day and night functional splint for patients with trapeziometacarpal osteoarthritis in improving pain and function

DETAILED DESCRIPTION:
Randomized clinical trial, and blind where selected 60 patients diagnosed with trapeziometacarpal osteoarthritis.Os patients were assessed by a blinded evaluator at the beginning of treatment and after 45, 90 and 180 days in relation to pain, thumb range of motion, strength hold, tweezers, dexterity, function and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients with osteoarthritis in accordance with the American College of Rheumatology classification criteria (ACR); of both genders and age above 18 years; Pain in TMC articulation between 3 and 8 cm in numerical pain scale (END) 10cm

Exclusion Criteria:

* Patients with severe deformities in hand with trapeziometacarpal osteoarthritis not possible to achieve pincer movement between the first, second and third fingers
* Deformity of the distal interphalangeal joint (IFD) of the thumb
* Use of splint the thumb in the last six months; Have surgery scheduled on hand for the next six months
* Allergy to the material of the splint
* Inability to respond to the questionnaire and perform the tests
* Geographic inaccessibility
* Infiltration in hand in the previous 3 months
* Changes in the use of anti-inflammatory and analgesic past 3 months
* Physiotherapy in hand over the last 3 months
* Have the following related diseases: carpal tunnel syndrome, carpal fractures of DeQuervain syndrome, tendonitis, fibromyalgia and chronic inflammatory arthropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Change in pain scale | baseline, after 45, 90 and 180 days

SECONDARY OUTCOMES:
Change in Functional capacity using the Cochin Hand Functional Scale questionnaire | baseline, after 45, 90 and 180 days
Change in pinch and grip strength | baseline, after 45, 90 and 180 days

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Sao Paulo - Rheumatology Division, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Silva FC, da Silva RVT, Meireles SM, Fernandes ADRC, Natour J. Daytime Functional Usage Versus Night-Time Wearing: Identifying the Optimal Wearing Regimen for a Custom-Made Orthosis in the Treatment of Trapeziometacarpal Osteoarthritis. Arch Phys Med Rehabil. 2024 Oct;105(10):1837-1845. doi: 10.1016/j.apmr.2024.06.013. Epub 2024 Jul 4. PMID 38971487